CLINICAL TRIAL: NCT06638164
Title: Evaluation of the Efficiency of Isolation Training Given to Caregivers of Isolated Individuals With Different Methods
Brief Title: Isolation Training Activity Given to Caregivers With Different Methods
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Beykent (Other)
Responsible Party: Principal Investigator, Hamiyet KIZIL, PhD RN Assistant Professor Hamiyet KIZIL, University of Beykent
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 12345
Record Dates: First submitted 2022-11-22; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Achievement; Knowledge; Satisfaction
Keywords: Isolation; Virtual Reality Glasses; Achievement; Knowledge; Satisfaction
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Experimental): No attempt was made to increase knowledge, skills and satisfaction. Standard procedure (oral explanation) was applied.
  Interventions: Other: Control
- Virtual Reality Glasses Group(Experiment) (Experimental): In order to increase knowledge, skills and satisfaction, isolation training was given with virtual reality glasses.
  Interventions: Other: Virtual reality glasses

INTERVENTIONS:
Other: Control — No attempt was made to increase knowledge, skills and satisfaction. Standard procedure (oral explanation) was applied.
  Arms: Control Group
Other: Virtual reality glasses — In order to increase knowledge, skills and satisfaction, isolation training was given with virtual reality glasses.
  Arms: Virtual Reality Glasses Group(Experiment)

SUMMARY:
The aim of this study; To measure the effectiveness of isolation training given to caregivers using different training methods. As a result of this measurement, the more effective method will be used routinely. In this way, it is aimed to create more conscious patients and caregivers. In this study, two different training methods will be used and the methods will be compared. Methods; It is divided into two as the experimental group, the training to be given with virtual glasses, and the training given with the control group, as the standard training booklet. With virtual glasses, patients will be trained in an interactive way with three-dimensional video, and they will be able to see and then apply them. The training to be given with the training booklet includes standard procedure and 2D visual and verbal expression. Based on this information, this study aims to evaluate the effectiveness of the Isolation Training Given to the Caregivers of Isolated Sick Individuals with Different Methods.

DETAILED DESCRIPTION:
This study was planned as a randomized controlled experimental study in order to evaluate the effectiveness of Isolation Training Given to Caregivers of Isolated Sick Individuals with Different Methods. The universe of the research will be the caregivers of the patients isolated in the intensive care and services of the Beykent University hospital, and the sample will be the caregivers of the patients whose hemodynamics are stable and willing to work. Sampling criteria; the patient's hemodynamics is stable, and the patients and their caregivers are willing to work. Power analysis was performed for the sample size of the study and it was decided to have a total of 60 patients, 30 in each group (control group, virtual reality group). Research data; structured information form, knowledge test for Isolation Measures, skills checklist for Isolation Measures and training satisfaction survey. Study data will be analyzed with SPSS 25 statistical program.

In the research; Two different training methods will be used and these are; Virtual Glasses application, which is the experimental group; For the care and follow-up of the isolated patient, a video will be taken and watched in order to show the caregivers that the personal protective equipment is worn correctly and in order, and this is explained. This video will be rendered 3D and shown to caregivers. Afterwards, the caregiver will be expected to apply the training received. The Control Group, on the other hand, will be trained with a training booklet to be applied as a standard procedure, which provides information on isolation methods.Before these trainings, knowledge test (pretest) and after training knowledge tests (posttest) will be done. During the training, the equipment will be worn by the caregivers, and the actions that are done / not done will be evaluated by marking from the checklist prepared during this process. Finally, the satisfaction with education questionnaire will be filled.With this study, it will be ensured that the Efficiency of the Isolation Training Given to the Caregivers of Isolated Sick Individuals with Different Methods.

ELIGIBILITY:
Inclusion Criteria:

The caregiver;

* The patient has a hospital infection that requires isolation,
* The patient has immune deficiency and the implementation of isolation measures,
* Not visually impaired
* Being able to read and write
* Written and verbal consent is obtained for participation in the study.

Exclusion Criteria:

The caregiver;

* The patient does not have a hospital infection that needs to be isolated,
* The patient has immune deficiency and isolation measures are not applied,
* Having a visually impaired being illiterate
* Written and verbal consent is not obtained for participation in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Achievement levels | 2 Months
  The caregivers of the isolated individuals were informed about the isolation precautions checklist.It was created in line with the literature to determine the knowledge levels regarding the ability to apply Isolation Precautions.It is a checklist consisting of 20 items that evaluates isolation precautions and wearing protective equipment, created by researchers in line with the literature. The lowest score that can be obtained from the checklist is "0", and the highest score is "100".
Knowledge levels | 2 Month
  The caregivers of the isolated individuals were informed about the knowledge exam.It is a survey consisting of 20 questions covering isolation precautions created by researchers in line with the literature.The lowest score that can be obtained from the knowledge exam is "0", and the highest score is "100".

SECONDARY OUTCOMES:
Satisfaction levels | 2 Months
  The caregivers of the isolated individuals were informed about the satisfaction with education questionnaire.The survey consists of 16 propositions. Each proposition is scored according to a 5-point Likert scale (1-strongly disagree, 2-disagree, 3-undecided, 4-agree, 5-strongly agree). It is determined that as the average scale score increases, individuals' satisfaction with the education method increases, and as the average scale score decreases, their satisfaction with the education method decreases. In the scale evaluation, individuals are given a minimum of 16 and a maximum of 80 points for their satisfaction with the education methods.

CONTACTS AND LOCATIONS:
Overall Officials: Hamiyet Kızıl, PhD RN, Principal Investigator — Beykent University; Hamiyet Kızıl, Principal Investigator — Beykent University
Locations (1):
- Beykent University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Butt, A. L., Kardong-Edgren, S., & Ellertson, A. (2018). Using game-based virtual reality with haptics for skill acquisition. Clinical Simulation in Nursing, 16, 25-32.
- [Result] Onturk ZK, Ugur E, Kocatepe V, Ates E, Ocaktan N, Unver V, Karabacak U. Use of simulation from high fidelity to low fidelity in teaching of safe-medication practices. J Pak Med Assoc. 2019 Feb;69(2):195-200. PMID 30804583
- [Result] Kolbe L, Jaywant A, Gupta A, Vanderlind WM, Jabbour G. Use of virtual reality in the inpatient rehabilitation of COVID-19 patients. Gen Hosp Psychiatry. 2021 Jul-Aug;71:76-81. doi: 10.1016/j.genhosppsych.2021.04.008. Epub 2021 Apr 29. PMID 33964789
- [Derived] Kizil H, Altintop I. Evaluation of the effectiveness of isolation training given to the caregivers of patients in isolation with different methods: a randomized controlled study. BMC Nurs. 2025 Sep 29;24(1):1219. doi: 10.1186/s12912-025-03662-0. PMID 41023681